CLINICAL TRIAL: NCT04721704
Title: Comparison of Efficacy and Safety of Triple Regimen Based on Clarithromycin VS Metronidazole in Pediatric Population in Pakistan
Brief Title: Comparison of Efficacy of Triple Regimen Based on Clarithromycin VS Metronidazole in Children
Acronym: CETR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shaheed Zulfiqar Ali Bhutto Medical University (Other)
Responsible Party: Principal Investigator, Dr.Nadia waheed, Assistant professor, Shaheed Zulfiqar Ali Bhutto Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: F-.1-1/2015/ERB/SZABMU/646
Record Dates: First submitted 2021-01-16; First posted 2021-01-25 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: H Pylori Gastritis
Keywords: H-pylori gastritis, eradication therapy, triple regimen
MeSH Terms: interventions — Omeprazole; Clarithromycin; Amoxicillin; Metronidazole

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Experimental): Group A will be given Amoxicillin AMO + Clarithromycin CLA + Proton pump inhibitor PPI based triple regimen
  Interventions: Drug: Clarithromycin+ Amoxicillin + Omeprazole
- Group B (Experimental): Group B will be given Amoxicillin AMO+ Metronidazole MET+ Proton pump inhibitor PPI based triple regimen
  Interventions: Drug: Metronidazole +Amoxicillin + Omeprazole

INTERVENTIONS:
Drug: Clarithromycin+ Amoxicillin + Omeprazole — In Group A: Amoxicillin AMO + Clarithromycin CLA + Proton pump inhibitor PPI will be given to children
  Other Names: Klaricid + Amoxil + Risek
  Arms: Group A
Drug: Metronidazole +Amoxicillin + Omeprazole — Group B: Amoxicillin AMO+ Metronidazole MET+ Proton pump inhibitor PPI
  Other Names: Flagyl + Amoxil + Risek
  Arms: Group B

SUMMARY:
All children from 1day to 18years of age, diagnosed with peptic ulcer disease due to H pylori at Pakistan Institute of Medical Sciences, Islamabad, from July 2020 to December 2021 will be included in the study. After informed written consent from parents/ guardians patients' bio data along with history and examination will be recorded on a proforma. They will be allocated into two groups, group A and group B randomly based on treatment regimen offered.

Group A: Amoxicillin AMO + Clarithromycin CLA + Proton pump inhibitor PPI) Group B: Amoxicillin AMO+ Metronidazole MET+ Proton pump inhibitor PPI The history will include presenting symptoms along duration, remission of symptoms after therapy and clinical outcome will also be recorded.

DETAILED DESCRIPTION:
Helicobacter pylori is a gram-negative bacillus responsible for one of the most common infections found in humans worldwide1. In general, the prevalence is high in developing countries and the infection is acquired at a young age. Most children infected with H pylori are asymptomatic. Antral gastritis is the most common manifestation in children. Duodenal and gastric ulcers may be associated with H pylori gastritis in 1.8 % children2. Antibiotic resistance is the major cause of failure in the treatment of H pylori infection3. Most of the studies worldwide confirmed an increase in macrolide resistance, while metronidazole resistance either decreased or remained stable. In a prospective multicenter European study, primarily comprised of adults, found a 31.8% resistance rate to clarithromycin and 25.7% to metronidazole in the study4.

If the strain is resistant to one of the antibiotics used, treatment success will be compromised5. As a result therapies that are recommended should be based on antibiotic susceptibility testing. If this testing is not available, then clarithromycin-based triple therapy should not be used as part of first-line therapy due to high rates of clarithromycin resistance rates6 The European Society for Paeditric Gastroenterology Hepatology and Nutrition/North American Society for Pediatric Gastroenterology, Hepatology and Nutrition made the recommendations in 2017 for the Management of Helicobacter pylori in Children that antimicrobial sensitivity should be obtained for the infecting H pylori to tailor eradication therapy accordingly and the effectiveness of first-line therapy should be evaluated in national/regional centers7.

If the strain is susceptible to clarithromycin (CLA) and to metronidazole (MET), triple therapy (PPI, amoxicillin [AMO], CLA) for 14 days and doses of proton pump inhibitor and antibiotics should be calculated based on the bodyweight8.

We aim to study efficacy and safety of clarithromycin vs metronidazole based triple regimen for the eradication of H pylori in children with peptic ulcer disease.

ELIGIBILITY:
Inclusion Criteria:

* 1. All children age 1-12 years having H-pylori gastritis

Exclusion Criteria:

* drug induced gastritis critically ill child

Ages: 1 Year to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Estimated)
Dates: Start 2020-09-14 (Actual); Primary Completion 2022-09-14 (Estimated); Study Completion 2022-09-14 (Estimated)

PRIMARY OUTCOMES:
Efficacy of Clarithromycin vs Metronidazole based triple regimen in treatment of H-pylori in induced Acid peptic disease in children in terms of reduction in duration of symptoms and negative Stool H-Pylori-Ag | 2 weeks
  All children age 1-12 years diagnosed with acid peptic disease with positive H-pylori Ag in stool will be randomized in to Group A & Group B and will be given either CLA or MET based triple eradication regimen. After 4 weeks of complication of triple regimen patients form both groups will be re-tested for H-pylori Ag in stool. The efficacy of both regimen will be compare in terms of duration of resolution of symptoms of Acid peptic disease and number of patients having negative stool H pylori Ag post treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Nadia Waheed, Principal Investigator — PIMS, SZABMU,ISLAMABAD
Locations (2):
- Pakistan (2):
  - Pakistan Institute of Medical Sciences,SZABMU, Islamabad, Capital Territory
  - Pakistan Institute of Medical Sciences, Islamabad, Islamabad, Islamabad

IPD SHARING:
Plan to Share IPD: Yes
SPSS DATA SHEETS WILL BE SHARED
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 6 months after publication for further 6 months
Access Criteria: through email on demand